CLINICAL TRIAL: NCT01499615
Title: A Prospective Study of a New Non-Invasive Cardiac Output Monitor in Children Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles Cote, Director of Clinical Research, Divisionof Pediatric Anesthesia, Massachusetts General Hospital
Other Study IDs: 2010-P-002709/1; MGH
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Children Receiving General Anesthesia
Keywords: adverse events; adverse cardiovascular events; early warning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- children undergoing general anesthesia: The intervention was the application of 4 ekg electrodes so as to non-invasivly measure cardiac output
  Interventions: Device: cardiac monitor

INTERVENTIONS:
Device: cardiac monitor — All children receive the same intervention which is the application of the 4 ekg electrodes

SUMMARY:
Traditionally cardiac output has been estimated with thermodilution. Recently a new non-invasive device has been approved by the FDA for use in children of all ages including neonates (just 4 EKG electrodes). Primary outcome: To prospectively collect simultaneous physiologic data for all enrolled children by transferring the data from the investigators computerized anesthesia records to Excel spreadsheets and to correlate adverse events across monitoring devices.

Secondary outcomes: To determine if the device provides meaningful data in terms of an early warning of decreased cardiac output in specific subgroups of children undergoing surgery and anesthesia, e.g., neonates, trauma patients, children with congenital heart disease, those undergoing procedures with expected blood loss, those undergoing laparoscopic procedures where gas insufflation may impede venous return to the heart.

DETAILED DESCRIPTION:
All children undergoing both elective and emergent surgery or GI endoscopy evaluation will be candidates for study. Since this is an FDA approved monitor that is approved across all age groups and since this is an additional monitor over those routinely used in the operating room and since it is noninvasive (4 EKG leads) verbal consent documented in the record has been approved by the IRB.

After informed verbal consent, either the research coordinator or a study physician will populate the cardiac output device with the child's age, weight, gender and height. For older children the required 4 EKG electrodes will be applied prior to induction of anesthesia (2 on the left side of the neck and 2 on the left chest at the level of the sternal depression; for neonates and infants one electrode can be applied to the forehead and the other to a thigh if application space is a problem). For children who are not able to be cooperative, as with most of our monitors the electrodes will be placed after induction of general anesthesia. An automated anesthesia record will continuously record heart rate, respiratory rate, oxygen saturation, systolic and diastolic pressures. The monitor will be set to perform these measurements every 1 minute. New software has been written that enables us to interface the cardiac output device with our automated anesthesia record. Thus the data from the cardiac output device will be inserted on the anesthesia record at approximate 1 minute intervals in real time. The data from the anesthesia records will later be downloaded as a unit to Excel spread sheets for later analysis. All demographic data will also be downloaded (age, weight, ASA physical status,surgical procedure) as well as blood loss and blood and fluid administered as well as drugs,significant intraoperative events, and the timing of events as they evolve. All data will be entered on a Partners password protected computer. Initially the patient's medical record number which links us to the electronic anesthesia record will be recorded as this allows us to download the data. Patient names will not be downloaded. Once the data set is completed,analyzed and locked, the medical record number will be removed so that no identifiers will remain. The data will not be shared with any other institution. Only deidentified data will remain on the final data base

ELIGIBILITY:
Inclusion Criteria:

* All children presenting to our operating rooms for general anesthesia

Exclusion Criteria:

* Cardiac surgery, open chest procedures

Ages: 1 Hour to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: neonates to teenagers
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Correlate adverse cardiovascular events in children under anesthesia with the cardiac output device and standard anesthesia monitors | approximately 18 months
  We plan to record all physiologic data from approximately 400 children under anesthesia and correlate adverse cardiovascular events determined by this new cardiac output device with standard anesthesia monitors

SECONDARY OUTCOMES:
determine if this device provides additonal safety for specific subgroups of pediatric patients under anesthesia e.g., those undergoing laparosopic procedures or procedures involving significant blood loss, neonates | approximatley 18 months
  determine is some subgroups within the proposed 400 cases derive specific benefit from this additional non-invasive monitor, i.e., an early warning of impaired cardiac output or a correlation with decreased blood pressure with decreased cardiac output. The issue is whether cardiac out updated at approximate 20 second intervals can provide an eralier warning than the standard 3 to 5 minute blood pressures provided by non-invasive blood pressure monitroing which is the standard of care.

CONTACTS AND LOCATIONS:
Locations (1):
- Operating rooms and GI endoscopy suites of the Massachusetts GeneralHospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] August DA, Sui J, Cote CJ. Unintentional epidural injection of 88 mug.kg(-1) of epinephrine. Paediatr Anaesth. 2014 Nov;24(11):1185-7. doi: 10.1111/pan.12503. Epub 2014 Aug 11. PMID 25130947
- [Derived] Cote CJ, Sui J, Anderson TA, Bhattacharya ST, Shank ES, Tuason PM, August DA, Zibaitis A, Firth PG, Fuzaylov G, Leeman MR, Mai CL, Roberts JD Jr. Continuous noninvasive cardiac output in children: is this the next generation of operating room monitors? Initial experience in 402 pediatric patients. Paediatr Anaesth. 2015 Feb;25(2):150-9. doi: 10.1111/pan.12441. Epub 2014 Jun 10. PMID 24916144